CLINICAL TRIAL: NCT05197777
Title: Innovations in Pain Assessment and Treatment for Individuals With Musculoskeletal Disorders: Brazil and Canada Collaboration
Brief Title: Pain Evaluation and Treatment in Clinical Settings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rubens da Silva (Other)
Collaborators: Londrina Santa casa Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Rubens da Silva, Professor, Université du Québec à Chicoutimi
Organization: Université du Québec à Chicoutimi (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 86.010-929
Record Dates: First submitted 2021-11-19; First posted 2022-01-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain; Functional Limitations; Musculoskeletal Disorders
Keywords: Pain; EEG; TMS
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Diseases; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 : conservator physiotherapy (Active Comparator): Education and exercices for pain relief by usual tradicional physiotherapy in Hospital: walking, mobility, and transfert.
  Interventions: Other: Conservative physiotherapy
- Group 2- tDCS associated to functional activities (Experimental): The intervention will start by a pretest on the first day (day 0, baseline record). Tdcs will be applied associated to physical task from functional activity of daily life. Functional task for the assessment of pain with high-tech tools for the implementation an experimental workstation, consisting in a hairdressing dummy head fixed to a telescopic table, adjustable to each individual's height. The dummy will be set at the height of the hands in a constrained position for the arms, i.e. with elbows flexed at 60 degrees. Elbow angles will be adjusted in a static position with a manual goniometer. The task will be performed in a standing position inside a 1m2 perimeter during 30 minutes. The elbow will be in a prolonged constraint position, undergoing repetitive movements, for 30 consecutive minutes. Performing a repetitive manual gesture. The cycle will be executed at a cadence of 30s/cycle with a metronome beat
  Interventions: Device: tDCS associated to functional activities

INTERVENTIONS:
Device: tDCS associated to functional activities — The intervention will start by a pretest on the first day (day 0, baseline record). Tdcs will be applied associated functional task from an experimental workstation, consisting in a hairdressing dummy head fixed to a telescopic table, adjustable to each individual's height. Elbow angles will be adjusted in a static position with a manual goniometer (60 degrees). The task will be performed in a standing position inside a 1m2 perimeter during 30 minutes, undergoing repetitive movements. Performing a repetitive manual gesture. The cycle will be executed at a cadence of 30s/cycle with a metronome beat. The TCT - tDCS Stimulator Kit Research version, with 35 cm2 on M1 of the contralateral hemisphere for the rigth dominant hand. During the first 30 s of active tDCS, an initial period of ''ramping up'' is administered, in which the stimulator reaches the maximum programmed current (2 mA) to mimic cutaneous perceptions. A 2 mA intensity will be maintained during activity.
  Arms: Group 2- tDCS associated to functional activities
Other: Conservative physiotherapy — Education and exercices for pain relief by usual tradicional physiotherapy in Hospital: walking, mobility, and transfert.
  Arms: Group 1 : conservator physiotherapy

SUMMARY:
This new research projet in pain is enrolled into an international official collaboration between researchers and clinicians from Irmandade da Santa Casa de Londrina (ISCAL) and those from two Quebec universities: University of Quebec in Chicoutimi (UQAC) and University of Quebec in Rimouski (UQAR).

ISCAL as a living laboratory research environment (sites, equipment, technology) for researchers, clinicians, students, and patients pool will make this project unique in the world, especially to stablish an integral concept on pain from identification, assessment and management, using neurophysiological central measures across patients with neuromusculoskeletal disorders. ISCAL in partnership with Santa Hospital in Londrina admit so many patients per day suffering of pain, by supporting a specific size of sample for establishment of this integral concept in pain.

This project builds on the foundations already well installed at ISCAL for data acquisition and storage, from an ideal set-up including patients with pain and clinicians. ISCAL infrastructure will be used to improve the acquirement of pain data from patients, using high-tech tools in a simple and robust experimental protocol targeting the central nervous system (CNS). Pain conventional evaluation (by questionnaires or simple questions related to pain intensity from anamneses or inspection doctor) will be completed by neurophysiological measures of the CNS activity based on the acquisition of biological signals and related to functional activities of the patients. A specific physiological behavior of pain will be determinate, using different types of preprocessing and statistical analyzes on biological signals. While pain and physical dysfunction mechanisms involve through the CNS, measurements from the CNS will allow to better understand the profiles and needs of the population (active adults and older people) suffering from pain and disabilities.

The knowledge acquired throughout this research program will improve the pain care in Santa Casa Hospital, the evidence-based practices (EBP) on site by specialist doctors and health professionals (nursing, medical, physiatry, physiotherapist etc.), and mainly will improve the quality of life of patients with pain. This project is a sharing of expertise beneficial to both poles, including the training of students, the use of advanced technologies and the exploration of new avenues in pain research grounded on the development of ISCAL in an international collaboration perspective.

All of the work from this research program aims to make ISCAL the reference center for chronic pain in Paraná (south of country) and further, for all Brazil.

DETAILED DESCRIPTION:
The purpose of this project is to detect pain and introduce an evaluation protocol and innovative therapeutic approach in the treatment of patients with chronic pain.

This project activities will be developed within the ISCAL structure, in five phases, as follows: Phase 1 - In this phase, it is aimed to determine the profile of patients admitted to the ISCAL outpatient clinic (pain profile, location of pain, age, gender, type of disorder, duration of symptoms, main functional limitations, type of work, among other variables), as well as, from meetings between the researchers, to establish a standardized pain assessment protocol using simple and high-tech measurement in different patients with musculoskeletal disorders; Phase 2 - This phase aims to determine the psychometric properties of biological measures of the central nervous system (such as parameters from electroencephalography and transcranial magnetic stimulation) in the context of neuromusculoskeletal pain. A secondary objective would also be to assess the validity (concurrent validity by correlations between measures), reliability (test-retest measure), and specificity of these measures; Phase 3 - In this phase, we aim to determine the sensitivity of pain detection measures from electroencephalography data and muscle fatigue (analyzed by electroneuromyography signals) in individuals with musculoskeletal disorders compared to age- and sex-matched controls. Phase 4 - In this phase, the objective is to verify the effect of pain management intervention using a combination of direct current stimulation neuromodulation (tDCS), transcutaneous electrical nerve stimulation (TENS) and transcranial magnetic stimulation (rTMS) protocols and other alternative pain management in individuals with musculoskeletal disorders. Finally in Phase 5, the objective is to provide subsidies for the creation of a research laboratory in pain, as well as possible workshops and lectures for the transfer of knowledge.

From this project, it is expected to contribute to a better knowledge of the mechanisms and neuromodulation of pain in the context of musculoskeletal disorders as well as to develop an evaluation protocol for these patients and help in future interventions or therapeutic options. Moreover, the use of validated assessment and treatment tools could represent an innovation in the rehabilitation context at ISCAL, and could bring benefits to the functionality and quality of life of patients with musculoskeletal disorders.

ELIGIBILITY:
Inclusion Criteria:

* Adults males and females
* Age ≥ 20 years and older (≤ 85)
* Body mass index (BMI) between 18 and 35 kg/m2
* From local the community, or be in the waiting list, or be admitted in ISCAL - Irmandande Santa Casa de Londrina (Londrina Santa Casa Hospital)
* Present, at least, 1 diagnosis of musculoskeletal disorder (medical diagnosis declared by the doctors of the clinical team of the hospital)
* Be able to present to the room and perform the tests and functional tasks, without and with minimal assistance
* Present a cognitive state greater than 20 in Mini-Mental State Examination.

Exclusion Criteria:

* Cancer
* Red flags (infection, tumor, etc.)
* Severe psychiatric disorders
* Palliative care
* Congenital spinal deformity (spondylolysis, intervertebral fusions, 4 lumbar vertebrae)
* Fairly severe systemic syndromes or diseases that may preclude testing
* Stroke - very acute phase (1 week) and this is until medial hemodynamic stability
* Any drugs or condition that could affect EEG or rMT measurements

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective and perception pain (score 1 to 10 numerical) | Change from baseline at 6 weeks
  The 0 (minimal) to 10 (maximal) numerical Rating Scales (NRS)
Subjective and perception pain (score total) | Change from baseline at 6 weeks
  Pain measurement using the Brain pain inventory (BPI) questionnaire. The interference items were now presented with 0-10 scales, with 0=no interference and 10=interferes completely
Objective pain by algometer (units in kgf) | Change from baseline at 6 weeks
  Algometer measurement for assessing the pressure pain threshold using a digital device in kgf.
Functional test #1 - The sitting-rising test (SRT; unit number of support from 10 to 1). | Change from baseline at 6 weeks
  he SRT basically consists in the quantification of the number of support (hands and/or knees, or hands or forearms on knees) one utilizes in order to sit and to rise from the floor. Independent grades are provided to each of the two actions - sitting and rising. The maximal grade is 5 for each one of the actions, losing one point for each support and additional half point for any detectable unbalance. The SRT allows, in very short time and practically in any place, the evaluation of many items - flexibility of lower limb joints, balance, motor coordination, and muscle power/body weight relationship - at the same time, which could be perhaps characterized as minimum functional muscular fitness.
Functional test #2 - Five Times Sit-to-Stand Test (Unit time in seconds) | Change from baseline at 6 weeks
  Assesses functional lower extremity strength, transitional movements, balance, and fall risk.Therapist Instructions: Have the patient sit with their back against the back of the chair. Count each stand aloud so that the patient remains oriented. Stop the test when the patient achieves the standing position on the 5th repetition.
  Patient Instructions: "Please stand up straight as quickly as you can 5 times, without stopping in between. Keep your arms folded across your chest. I'll be timing you with a stopwatch. Ready, begin
Functional test #3 Timed Up and Go test (TUG, unit time in seconds) | Change from baseline at 6 weeks
  Purpose: To assess mobility. Equipment: A stopwatch. Directions: Patients wear their regular footwear and can use a walking aid, if needed. Begin by having the patient sit back in a standard arm chair and identify a line 3 meters, or 10 feet away, on the floor.
Nordic Musculoskeletal Questionnaire (NMQ) | Change from baseline at 6 weeks
  The Nordic Musculoskeletal Questionnaire (NMQ) quantifies musculoskeletal pain and activity prevention in 9 body regions. The questionnaire can determine the prevalence of chronic pain across all participants. The NMQ is a self-administrated standardized questionnaire collecting sociodemographic information, health status, and musculosketal region pain.

SECONDARY OUTCOMES:
Muscle measurement by recording EMG signals (Units in microvolts μV) | Change from baseline at 6 weeks
  Muscular activity will be measured durinh physical function .e. under 30-minutes of an experimental functional task, time up and go test and a 6 meters walk test, using a wireless BTS FREEEMG 300
Brain measurement by recording EEG signals (Units in microvolts μV and frequency in Hz) | Change from baseline at 6 weeks
  Brain measurement by recording EEG signals at rest, during physical function i.e. under 30-minutes of an experimental functional task, time up and go test and a 6 meters walk test, using an Emotiv wireless EPOC® EEG Headset
Cortical excitability was assessed with the resting motor threshold (rMT) using a Transcranial Magnetic Stimulator (Units in microvolts μV) | Change from baseline at 6 weeks
  Transcranial Magnetic Stimulator (Magstim Company Ltd., UK). rMT was defined as the minimal intensity of stimulation capable of eliciting MEPs of at least 50 yV in 50% of the trials with the muscle at rest, expressed in percentage of the maximum stimulator output.
  rMT will be assessed at day 0 after 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Suzy Ngomo, PhD, Study Director — Université du Québec à Chicoutimi (UQAC); Hassan Ezzaidi, PhD, Study Chair — Université du Québec à Chicoutimi; Mohamed Bahoura, PhD, Study Chair — Université du Québec à Rimouski; Marcos Parron, PhD, Study Chair — ISCAL - Londrina Santa Casa Hospital; Fahd Fahd Haddad, MD, Study Chair — ISCAL - Londrina Santa casa Hospital; Colince Segning, MSc, Study Chair — Université du Québec à Chicoutimi
Locations (1):
- Karen Fernandes, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nordander C, Ohlsson K, Akesson I, Arvidsson I, Balogh I, Hansson GA, Stromberg U, Rittner R, Skerfving S. Risk of musculoskeletal disorders among females and males in repetitive/constrained work. Ergonomics. 2009 Oct;52(10):1226-39. doi: 10.1080/00140130903056071. PMID 19787502
- [Result] Mahdavi N, Motamedzade M, Jamshidi AA, Darvishi E, Moghimbeygi A, Heidari Moghadam R. Upper trapezius fatigue in carpet weaving: the impact of a repetitive task cycle. Int J Occup Saf Ergon. 2018 Mar;24(1):41-51. doi: 10.1080/10803548.2016.1234706. Epub 2016 Oct 6. PMID 27707416
- [Result] Srinivasan D, Mathiassen SE. Motor variability in occupational health and performance. Clin Biomech (Bristol). 2012 Dec;27(10):979-93. doi: 10.1016/j.clinbiomech.2012.08.007. Epub 2012 Sep 4. PMID 22954427
- [Result] Leboeuf-Yde C, Nielsen J, Kyvik KO, Fejer R, Hartvigsen J. Pain in the lumbar, thoracic or cervical regions: do age and gender matter? A population-based study of 34,902 Danish twins 20-71 years of age. BMC Musculoskelet Disord. 2009 Apr 20;10:39. doi: 10.1186/1471-2474-10-39. PMID 19379477
- [Result] Nasseroleslami B, Lakany H, Conway BA. EEG signatures of arm isometric exertions in preparation, planning and execution. Neuroimage. 2014 Apr 15;90:1-14. doi: 10.1016/j.neuroimage.2013.12.011. Epub 2013 Dec 16. PMID 24355482
- [Result] Neuper C, Wortz M, Pfurtscheller G. ERD/ERS patterns reflecting sensorimotor activation and deactivation. Prog Brain Res. 2006;159:211-22. doi: 10.1016/S0079-6123(06)59014-4. PMID 17071233
- [Result] Pfurtscheller G, Lopes da Silva FH. Event-related EEG/MEG synchronization and desynchronization: basic principles. Clin Neurophysiol. 1999 Nov;110(11):1842-57. doi: 10.1016/s1388-2457(99)00141-8. PMID 10576479
- [Result] Descatha A, Roquelaure Y, Chastang JF, Evanoff B, Melchior M, Mariot C, Ha C, Imbernon E, Goldberg M, Leclerc A. Validity of Nordic-style questionnaires in the surveillance of upper-limb work-related musculoskeletal disorders. Scand J Work Environ Health. 2007 Feb;33(1):58-65. doi: 10.5271/sjweh.1065. PMID 17353966
- [Result] Descatha A, Roquelaure Y, Chastang JF, Evanoff B, Cyr D, Leclerc A. Work, a prognosis factor for upper extremity musculoskeletal disorders? Occup Environ Med. 2009 May;66(5):351-2. doi: 10.1136/oem.2008.042630. No abstract available. PMID 19376942
- [Result] Karcioglu O, Topacoglu H, Dikme O, Dikme O. A systematic review of the pain scales in adults: Which to use? Am J Emerg Med. 2018 Apr;36(4):707-714. doi: 10.1016/j.ajem.2018.01.008. Epub 2018 Jan 6. PMID 29321111
- [Result] Maskeliunas R, Damasevicius R, Martisius I, Vasiljevas M. Consumer-grade EEG devices: are they usable for control tasks? PeerJ. 2016 Mar 22;4:e1746. doi: 10.7717/peerj.1746. eCollection 2016. PMID 27014511
- [Result] Wang D, Miao D, Blohm G. Multi-class motor imagery EEG decoding for brain-computer interfaces. Front Neurosci. 2012 Oct 9;6:151. doi: 10.3389/fnins.2012.00151. eCollection 2012. PMID 23087607
- [Result] Segning CM, Ezzaidi H, da Silva RA, Ngomo S. A Neurophysiological Pattern as a Precursor of Work-Related Musculoskeletal Disorders Using EEG Combined with EMG. Int J Environ Res Public Health. 2021 Feb 19;18(4):2001. doi: 10.3390/ijerph18042001. PMID 33669544
- [Result] Desbiens S, Girardin-Rondeau M, Guyot-Messier L, Lamoureux D, Paris L, da Silva RA, Ngomo S. Effect of transcranial direct stimulation combined with a functional task on fibromyalgia pain: A case study. Neurophysiol Clin. 2020 Apr;50(2):134-137. doi: 10.1016/j.neucli.2020.02.006. Epub 2020 Mar 20. No abstract available. PMID 32205006